CLINICAL TRIAL: NCT03838211
Title: tDCS-accompanied Cognitive Training Effects in Healthy Older Adults - Randomised, Sham Controlled, Interventional Study
Brief Title: Brain Stimulation and Cognitive Training in Healthy Older Adults
Acronym: TrainStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TrainStim3
Record Dates: First submitted 2019-02-01; First posted 2019-02-12 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Aging
Keywords: memory; brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stimulation group (Experimental): Anodal tDCS + intensive cognitive Training
  Interventions: Device: Anodal tDCS; Behavioral: Intensive cognitive training
- sham group (Sham Comparator): Sham tDCS + intensive cognitive Training
  Interventions: Behavioral: Intensive cognitive training

INTERVENTIONS:
Device: Anodal tDCS — Anodal transcranial direct current stimulation (tDCS), 9 sessions with 20 minutes stimulation each (current intensity of 1mA)
  Arms: stimulation group
Behavioral: Intensive cognitive training — Intensive cognitive training of a letter memory updating task and a 3-stage Markov decision making task, 9 sessions

SUMMARY:
The aim of this study is to investigate whether a tDCS-accompanied intensive cognitive training of working memory leads to performance improvement in healthy older individuals.

DETAILED DESCRIPTION:
The goal of the present study is to assess behavioral (primary) and neural effects of a multi-session cognitive training combined with transcranial direct current stimulation (tDCS). Many studies to date have found tDCS to be an efficient method to enhance various cognitive functions by modulating cortical excitability in young adults, but its behavioral impact and underlying mechanisms in aging still need to be elucidated. Healthy older adults will participate in a three-week cognitive training with concurrent online tDCS application. Cognitive performance (primary), as well as structural and functional imaging data will be examined before, during and after the intervention. In order to draw conclusions about the effect of tDCS in addition to cognitive training, a control group, receiving sham stimulation during training, will be assessed. Furthermore, to assess neural correlates of performance improvement, functional and structural parameters will be measured with MRI before and after training. Follow-up sessions to assess long-term effects are planned four weeks and six months after the post assessment. The results of the study will offer valuable insights into efficacy of combined tDCS and cognitive training, as compared to training alone, in older adults. Moreover, improved understanding of tDCS effects on cognitive training performance and underlying neural correlates may help to develop novel approaches for cognitive decline in healthy and pathological aging.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (65 - 80 years);
* Right handedness;
* Unobtrusive neuropsychological screening

Exclusion Criteria:

* Mild cognitive impairment (MCI) or dementia; other neurodegenerative neurological disorders; epilepsy; previous stroke;
* Severe and untreated medical conditions that precludes participation in the training, as determined by responsible physician;
* History of severe alcoholism or use of drugs;
* Severe psychiatric disorders such as depression (if not in remission) or psychosis;
* Contraindication for MRI (claustrophobia, metallic implants, ferromagnetic metals in the body, disorders of thermoregulation, pregnant women)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Working memory training performance (Letter Updating task) | 3 weeks
  Performance in a memory training task (Letter updating) under anodal tDCS compared to sham condition;operationalized by working Memory Updating performance assessed with number of correctly recalled letter lists in the letter updating task, analyzed immediately after training period (anodal condition versus sham)

SECONDARY OUTCOMES:
Working memory training performance (Markov task) | 3 weeks
  Performance in second memory training task (Markov decision making) under anodal tDCS compared to sham condition, analyzed immediately after training period (anodal condition versus sham)
Transfer outcomes | 3 weeks
  Performance in cognitive transfer tasks, comparing performance immediately before and after training period (anodal condition versus sham)
Long-term outcomes | 4 weeks after training, 6 months after 4-week follow-up
  Long-term performance in training and transfer tasks, comparing performance immediately before and after training period with performance at 4 weeks and 6-months after training period (anodal condition versus sham)
Neural correlates | 3 weeks, 6 months
  Structural and functional neural correlates of the intervention, as measured by structural, functional resting-state and diffusion weighted MRI, immediately before and after the intervention and 6 months after follow-up (anodal condition versus sham)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof., Study Director — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thams F, Li SC, Floel A, Antonenko D. Functional Connectivity and Microstructural Network Correlates of Interindividual Variability in Distinct Executive Functions of Healthy Older Adults. Neuroscience. 2023 Aug 21;526:61-73. doi: 10.1016/j.neuroscience.2023.06.005. Epub 2023 Jun 14. PMID 37321368
- [Derived] Antonenko D, Fromm AE, Thams F, Grittner U, Meinzer M, Floel A. Microstructural and functional plasticity following repeated brain stimulation during cognitive training in older adults. Nat Commun. 2023 Jun 2;14(1):3184. doi: 10.1038/s41467-023-38910-x. PMID 37268628
- [Derived] Antonenko D, Thams F, Uhrich J, Dix A, Thurm F, Li SC, Grittner U, Floel A. Effects of a Multi-Session Cognitive Training Combined With Brain Stimulation (TrainStim-Cog) on Age-Associated Cognitive Decline - Study Protocol for a Randomized Controlled Phase IIb (Monocenter) Trial. Front Aging Neurosci. 2019 Aug 16;11:200. doi: 10.3389/fnagi.2019.00200. eCollection 2019. PMID 31474848

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT03838211/SAP_000.pdf